CLINICAL TRIAL: NCT03188536
Title: Clinical and Sociodemographic Characterization of Multiple Myeloma Patients With Symptomatic Relapse and/or Refractory Disease in Spain
Brief Title: Clinical and Sociodemographic Characterization of Multiple Myeloma Participants With Symptomatic Relapse and/or Refractory Disease in Spain (CharisMMa Study)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: RRMM-5012; TAK-MMR-2017-01 (Registry Identifier: Spanish health authority)
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Myeloma (MM) Participants: Adult participants with a diagnosis of MM who received at least one previous treatment line (standard care of treatment) and experienced symptomatic relapse and/or refractory disease in the previous 6 months, who were followed-up at the time of the study visit. No intervention was administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As it was an observational study, no intervention was administered in this study.

SUMMARY:
The purpose of this study is to characterize the multiple myeloma (MM) participants with symptomatic relapse and/or refractory disease in Spain.

DETAILED DESCRIPTION:
Adult participants with a diagnosis of MM who have received at least one previous treatment line and have experienced symptomatic relapse and/or refractory disease in the previous 6 months, who are still in follow-up at the time of the study visit will be observed in this study.

The study will look into sociodemographic data, current clinical and therapeutic data, clinical data relative to the latest relapse and clinical data at diagnosis and previous relapses will be collected.

The study will enroll approximately 350 patients.

This multi-center trial will be conducted in a total of 30 public sites in Spain. The overall time to collect data will be approximately 1 year from June 2017 to May 2018.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of MM and has received at least one previous treatment line.
* Have experienced symptomatic relapse and/or refractory disease in the 6 months before the study.
* Has continued in follow-up at the time of the study visit.
* Is currently treated in the site who have clinical records available.
* Is capable of understanding and completing the questions in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), and EORTC Multiple Myeloma Module (QLQ-MY20) questionnaires.

Exclusion Criteria:

• Participants who do not agree to participate in the study or who do not give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of MM who have received at least one previous treatment line and have experienced symptomatic relapse and/or refractory disease in the previous 6 months, who are still in follow-up at the time of the study visit will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Science, Study Director — Takeda
Locations (30):
- Spain (30):
  - H Universitario Puerta del Mar, Cadiz, Andalusia
  - H Virgen de las Nieves, Granada, Andalusia
  - Hospital Juan Ramon Jimenez, Huelva, Andalusia
  - H Jerez, Jerez de la Frontera, Andalusia
  - Hospital Costa del Sol, Marbella, Andalusia
  - H. Nuestra Senora de Valme, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - H Son Espases, Palma, Balearic Islands
  - Hospital Son Llatzer, Palma, Balearic Islands
  - H de Donosti, Donostia / San Sebastian, Basque Country
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Basque Country
  - H U Canarias, San Cristóbal de La Laguna, Canary Islands
  - H Marques de Valdecilla, Santander, Cantabria
  - Hospital de Burgos, Burgos, Castille and León
  - Hospital de Leon, León, Castille and León
  - Hospital de Salamanca, Salamanca, Castille and León
  - Complejo Asistencial de Segovia, Segovia, Castille and León
  - H U de Guadalajara, Guadalajara, Castille-La Mancha
  - Complejo Hospitalario Toledo, Toledo, Castille-La Mancha
  - Hospital Clinico de Barcelona, Barcelona, Catalonia
  - Hospital Doctor Trueta ICO Girona, Girona, Catalonia
  - ICO Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - H Universitari de Tarragona Joan XXIII, Tarragona, Catalonia
  - Hospital Lucus Agusti, Lugo, Galicia
  - H Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - H Universitario de Cabuenes, Gijón, Principality of Asturias
  - H Infanta Leonor, Madrid
  - H 12 de Octubre, Madrid
  - H Clinico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Dachs LR, Gaisan CM, Bustamante G, Lopez SG, Garcia EG, Persona EP, Gonzalez-Calle V, Auzmendi MS, Perez JMA, Gonzalez Montes Y, Rios Tamayo R, de Miguel Llorente D, Bernal LP, Mayol AS, Caro CC, Grande M, Fernandez-Nistal A, Naves A, Miguel EMOS. Assessment of the psychometric properties of the Spanish version of EORTC QLQ-MY20 and evaluation of health-related quality of Life outcomes in patients with relapsed and/or refractory multiple myeloma in the real-world setting in Spain: results from the CharisMMa study. Leuk Lymphoma. 2023 Nov-Dec;64(11):1847-1856. doi: 10.1080/10428194.2023.2240922. Epub 2023 Aug 4. PMID 37539698
- [Derived] Ocio EM, Montes-Gaisan C, Bustamante G, Garzon S, Gonzalez E, Perez-Persona E, Gonzalez-Calle V, Sirvent M, Arguinano JM, Gonzalez Y, Rios R, de Miguel D, Grande M, Fernandez-Nistal A, Naves A, Rosinol L. Real-World Health Care Services Utilization Associated With the Management of Patients With Relapsed and Refractory Multiple Myeloma in Spain: The CharisMMa Study. Clin Lymphoma Myeloma Leuk. 2023 Oct;23(10):e341-e347. doi: 10.1016/j.clml.2023.07.006. Epub 2023 Jul 15. PMID 37517875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in Spain from 26 July 2017 to 30 January 2019.
Pre-assignment Details: Participants with a diagnosis of multiple myeloma with symptomatic relapse and/or refractory disease were observed to collect the retrospective data on Day 1.
Groups:
- Multiple Myeloma (MM) Participants: Adult participants with a diagnosis of MM received at least one previous treatment line (standard care of treatment) and experienced symptomatic relapse and/or refractory disease in the previous 6 months, who were followed-up at the time of the study visit. No intervention was administered in this study.
Period: Overall Study
Arm/Group | Multiple Myeloma (MM) Participants
Started | 282
Completed | 276
Not Completed | 6
Not completed — No relapse/refractoriness(last 6 months) | 5
Not completed — Not participated/met inclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: All participants eligible for analyses were included.
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 147
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 276
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI=Weight (kg)/Height(m)^2.
  Kg/m^2 | 27.5 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of MM Participants Categorized by Sociodemographic Variables at Diagnosis
Description: Sociodemographic variables included age(in years), sex(male or female), body mass index(BMI), residence(rural or urban), educational level(illiterate,no studies(can only read/write),primary studies,secondary studies,higher studies), work status(unemployed,active employment,temporarily/ permanently disabled, retired, other), cohabitation(lives-alone,with relatives,alone with help from a caregiver), need for financial assistance (yes/no), degree of dependence(independent,dependent:grade I-requires help to perform activities of daily living [ADL] at least once a day,grade II-needs help to perform ADLs 2 or 3 times a day or grade III-needs help to perform ADLs several times a day), healthy habits (high[jogging;climbing;cycling;swimming;sports;intensive work;moving >20 kg loads], moderate[walking;dancing;domestic chores;sports with children,walking house pets;general construction work;moving <20 kg loads] physical activity or inactive, smoking habit (yes/no), alcohol use (yes/no).
Time Frame: Day 1
Population: All participants eligible for analyses were included. Number analyzed is the number of participants with data available for analyses for the specific category. Percentages were rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
percentage of participants
  Age, Adults (27-90 years) | 100
  Sex, Male | 53.3
  Sex, Female | 46.7
  BMI, 15 to 52 kg/m^2 | 100
  Area of Residence, Rural | 24.3
  Area of Residence, Urban | 75.7
  Educational level, Illiteracy: number analyzed (Participants) | 270
  Educational level, Illiteracy | 0.7
  Educational level, No Studies (just read/write): number analyzed (Participants) | 270
  Educational level, No Studies (just read/write) | 10.4
  Educational level, Primary studies: number analyzed (Participants) | 270
  Educational level, Primary studies | 43.3
  Educational level, Secondary studies: number analyzed (Participants) | 270
  Educational level, Secondary studies | 34.1
  Educational level, Higher studies: number analyzed (Participants) | 270
  Educational level, Higher studies | 11.5
  Work Status, Unemployed: number analyzed (Participants) | 275
  Work Status, Unemployed | 5.5
  Work Status, Active: number analyzed (Participants) | 275
  Work Status, Active | 5.1
  Work Status, Temporary/permanent disability: number analyzed (Participants) | 275
  Work Status, Temporary/permanent disability | 20.0
  Work Status, Retired: number analyzed (Participants) | 275
  Work Status, Retired | 65.1
  Work Status, Other: number analyzed (Participants) | 275
  Work Status, Other | 4.4
  Cohabitation status, Living Alone: number analyzed (Participants) | 274
  Cohabitation status, Living Alone | 12.4
  Cohabitation status, Living with Relatives: number analyzed (Participants) | 274
  Cohabitation status, Living with Relatives | 85.8
  Cohabitation, Living Alone with Assistance: number analyzed (Participants) | 274
  Cohabitation, Living Alone with Assistance | 1.8
  Need of Financial Support, No: number analyzed (Participants) | 274
  Need of Financial Support, No | 93.8
  Level of Dependence, Independent: number analyzed (Participants) | 275
  Level of Dependence, Independent | 71.3
  Level of Dependence, Grade I: number analyzed (Participants) | 275
  Level of Dependence, Grade I | 14.5
  Level of Dependence, Grade II: number analyzed (Participants) | 275
  Level of Dependence, Grade II | 12.7
  Level of Dependence, Grade III: number analyzed (Participants) | 275
  Level of Dependence, Grade III | 1.5
  Physical Activity, High: number analyzed (Participants) | 275
  Physical Activity, High | 1.8
  Physical Activity, Moderate: number analyzed (Participants) | 275
  Physical Activity, Moderate | 45.8
  Physical Activity, Inactive: number analyzed (Participants) | 275
  Physical Activity, Inactive | 52.4
  Current smoking habit, Yes | 3.6
  Current smoking habit, No | 96.4
  Alcohol Use, Yes | 6.5
  Alcohol Use, No | 93.5

2. Primary Outcome: Percentage of MM Participants Categorized by Clinical Variables at Diagnosis
Description: Clinical variables at Diagnosis included age,MM type(heavy/light chain/Bence-Jones protein), international staging system(ISS),disease stage(I:low risk,β2-Microglobulin<3.5mg/L and albumin≥3.5g/dL,II:not stage I or III,III:high risk,β2-Microglobulin≥5.5mg/L),calcium,renal insufficiency,anemia or bone lesions(CRAB) signs(serum calcium>0.25mmol/L upper limit of normal,renal failure-creatinine clearance<40mL/min/serum creatinine>117μmol/L, anemia:reduction of hemoglobin(Hb)>2g/dL below lower limit of normal or Hb<10g/dL,bone lesions 1/more osteolytic lesion,cytogenetic abnormalities(t[4;14],t[11;14],t[14;16],t[14;20],t[6;14],trisomies,d[17p],g[1q]/others), risk according to cytogenetic profile(standard:trisomies,t[11;14];t[6;14],intermediate:t[4;14],g[1q], high:d[17p],t[14;16],t[14;20],other), eastern cooperative oncology group(ECOG) status (0:fully active,1:restricted physical activity,2:ambulatory,unable to carry out any work,3:capable of limited selfcare,4:completely disabled,5:dead).
Time Frame: Day 1
Population: All participants eligible for analyses were included. Number analyzed is the number of participants with data available for analyses for the specific category. Participants are repeated for multiple CRAB signs and cytogenic abnormalities. Percentages were rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
percentage of participants
  Age, Adults (27-90 years) | 100
  MM Type, Heavy chain, IgA: number analyzed (Participants) | 266
  MM Type, Heavy chain, IgA | 24.1
  MM Type, Heavy chain, IgD: number analyzed (Participants) | 266
  MM Type, Heavy chain, IgD | 1.9
  MM Type, Heavy chain, IgG: number analyzed (Participants) | 266
  MM Type, Heavy chain, IgG | 56.8
  MM Type, Heavy chain, IgM: number analyzed (Participants) | 266
  MM Type, Heavy chain, IgM | 0.8
  MM Type, Heavy chain, No Heavy Chain: number analyzed (Participants) | 266
  MM Type, Heavy chain, No Heavy Chain | 16.5
  MM Type, Light Chain, No Light Chain | 3.3
  MM Type, Light Chain, Kappa | 59.8
  MM Type, Light Chain, Lambda | 37.0
  MM Type, Bence Jones Protein, Yes: number analyzed (Participants) | 235
  MM Type, Bence Jones Protein, Yes | 53.6
  ISS Disease Stage I: number analyzed (Participants) | 267
  ISS Disease Stage I | 28.8
  ISS Disease Stage II: number analyzed (Participants) | 267
  ISS Disease Stage II | 28.1
  ISS Disease Stage III: number analyzed (Participants) | 267
  ISS Disease Stage III | 43.1
  CRAB Signs, None | 12.7
  CRAB Signs, Some, Increase in blood calcium levels: number analyzed (Participants) | 241
  CRAB Signs, Some, Increase in blood calcium levels | 12.0
  CRAB Signs, Some, Renal failure: number analyzed (Participants) | 241
  CRAB Signs, Some, Renal failure | 18.7
  CRAB Signs, Some, Anemia: number analyzed (Participants) | 241
  CRAB Signs, Some, Anemia | 52.7
  CRAB Signs, Some, Bone lesions: number analyzed (Participants) | 241
  CRAB Signs, Some, Bone lesions | 76.3
  Cytogenetic abnormalities, t (4;14): number analyzed (Participants) | 106
  Cytogenetic abnormalities, t (4;14) | 11.3
  Cytogenetic abnormalities, t (11;14): number analyzed (Participants) | 106
  Cytogenetic abnormalities, t (11;14) | 14.2
  Cytogenetic abnormalities, t (14;16): number analyzed (Participants) | 106
  Cytogenetic abnormalities, t (14;16) | 1.9
  Cytogenetic abnormalities, Trisomies: number analyzed (Participants) | 106
  Cytogenetic abnormalities, Trisomies | 3.8
  Cytogenetic abnormalities, d (17p): number analyzed (Participants) | 106
  Cytogenetic abnormalities, d (17p) | 17.9
  Cytogenetic abnormalities, g (1q): number analyzed (Participants) | 106
  Cytogenetic abnormalities, g (1q) | 21.7
  Cytogenetic abnormalities, Other: number analyzed (Participants) | 106
  Cytogenetic abnormalities, Other | 66.0
  Risk, High: number analyzed (Participants) | 106
  Risk, High | 19.8
  Risk, Standard: number analyzed (Participants) | 106
  Risk, Standard | 12.3
  Risk, Intermediate: number analyzed (Participants) | 106
  Risk, Intermediate | 23.6
  Risk, Other: number analyzed (Participants) | 106
  Risk, Other | 44.3
  ECOG Status, 0: number analyzed (Participants) | 195
  ECOG Status, 0 | 29.7
  ECOG Status, 1: number analyzed (Participants) | 195
  ECOG Status, 1 | 41.5
  ECOG Status, 2: number analyzed (Participants) | 195
  ECOG Status, 2 | 22.6
  ECOG Status, 3: number analyzed (Participants) | 195
  ECOG Status, 3 | 6.2

3. Primary Outcome: Percentage of MM Participants Categorized by Clinical Variables at Latest Symptomatic Relapse and/or Refractory Episode
Description: Clinical variables include date of latest symptomatic relapse and/or refractory episode, ISS disease stage, CRAB signs, other clinical variables (plasmacytomas: medullary or extramedullary, diffuse osteopenia, fractures, neurological symptoms, infections, concomitant diseases like diabetes, neuropathy, chronic obstructive pulmonary disease (COPD), cardiovascular disease, liver failure, psychiatric and/or neurological disorders, any other secondary disorders, cytogenetic abnormalities, risk according to cytogenetic profile at relapse(standard:trisomies,t[11;14];t[6;14],intermediate:t[4;14],g[1q], high:d[17p],t[14;16],t[14;20],other), treatment started after latest symptomatic relapse and/or refractory episode.
Time Frame: Day 1
Population: All participants eligible for analyses were included. Number analyzed is the number of participants with data available for analyses for the specific category. Participants are repeated across multiple categories. Percentages were rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
percentage of participants
  Relapse Within 6 Months of Last Relapse | 61.6
  ISS Disease Stage I: number analyzed (Participants) | 211
  ISS Disease Stage I | 37.4
  ISS Disease Stage II: number analyzed (Participants) | 211
  ISS Disease Stage II | 35.5
  ISS Disease Stage III: number analyzed (Participants) | 211
  ISS Disease Stage III | 27.0
  CRAB Signs, None | 25.7
  CRAB Signs, Some-Increase in blood calcium levels: number analyzed (Participants) | 205
  CRAB Signs, Some-Increase in blood calcium levels | 9.3
  CRAB Signs, Some-Renal Failure: number analyzed (Participants) | 205
  CRAB Signs, Some-Renal Failure | 20.5
  CRAB Signs, Some-Anemia: number analyzed (Participants) | 205
  CRAB Signs, Some-Anemia | 43.9
  CRAB Signs, Some-Bone lesions: number analyzed (Participants) | 205
  CRAB Signs, Some-Bone lesions | 65.9
  Cytogenetic Abnormalities, t(4;14): number analyzed (Participants) | 87
  Cytogenetic Abnormalities, t(4;14) | 11.5
  Cytogenetic Abnormalities, t(11;14): number analyzed (Participants) | 87
  Cytogenetic Abnormalities, t(11;14) | 8.0
  Cytogenetic Abnormalities, t(14;16): number analyzed (Participants) | 87
  Cytogenetic Abnormalities, t(14;16) | 5.7
  Cytogenetic Abnormalities, Trisomies: number analyzed (Participants) | 87
  Cytogenetic Abnormalities, Trisomies | 4.6
  Cytogenetic Abnormalities, d (17p): number analyzed (Participants) | 87
  Cytogenetic Abnormalities, d (17p) | 19.5
  Cytogenetic Abnormalities, g (1q): number analyzed (Participants) | 87
  Cytogenetic Abnormalities, g (1q) | 27.96
  Cytogenetic Abnormalities, other: number analyzed (Participants) | 87
  Cytogenetic Abnormalities, other | 64.4
  Risk, High: number analyzed (Participants) | 49
  Risk, High | 38.8
  Risk, Standard: number analyzed (Participants) | 49
  Risk, Standard | 12.2
  Risk, Intermediate: number analyzed (Participants) | 49
  Risk, Intermediate | 49.0
  Diffuse osteopathy: number analyzed (Participants) | 272
  Diffuse osteopathy | 15.4
  Fractures | 15.2
  Neurological symptoms | 8.0
  Infections | 15.2
  Comorbidities, Diabetes: number analyzed (Participants) | 175
  Comorbidities, Diabetes | 24.6
  Comorbidities, Neuropathy: number analyzed (Participants) | 175
  Comorbidities, Neuropathy | 20.6
  Comorbidities, Nephropathy: number analyzed (Participants) | 175
  Comorbidities, Nephropathy | 15.4
  Comorbidity, COPD: number analyzed (Participants) | 175
  Comorbidity, COPD | 11.4
  Comorbidities, Cardiovascular disease: number analyzed (Participants) | 175
  Comorbidities, Cardiovascular disease | 48.6
  Comorbidities, Liver failure: number analyzed (Participants) | 175
  Comorbidities, Liver failure | 1.7
  Comorbidities,Psychiatric or Neurological Disorder: number analyzed (Participants) | 175
  Comorbidities,Psychiatric or Neurological Disorder | 14.3
  Comorbidities, Other secondary disorders: number analyzed (Participants) | 175
  Comorbidities, Other secondary disorders | 45.7
  Medullary Plasmacytoma | 15.3
  Extramedullary Plasmacytoma | 15.6
  Anti-CD38 mAb Monotherapy, Second Line: number analyzed (Participants) | 112
  Anti-CD38 mAb Monotherapy, Second Line | 0.9
  Anti-CD38 mAb Monotherapy, Third Line: number analyzed (Participants) | 68
  Anti-CD38 mAb Monotherapy, Third Line | 13.2
  Anti-CD38 mAb Monotherapy, Fourth Line or Later: number analyzed (Participants) | 79
  Anti-CD38 mAb Monotherapy, Fourth Line or Later | 20.3
  Double PI Therapy+Steroids/Alkylating Agent,2 Line: number analyzed (Participants) | 112
  Double PI Therapy+Steroids/Alkylating Agent,2 Line | 9.8
  Double PI therapy+Steroids/Alkylating Agent,3 Line: number analyzed (Participants) | 68
  Double PI therapy+Steroids/Alkylating Agent,3 Line | 10.3
  DoublePI Therapy+Steroids/Alkylating Agent,>=4Line: number analyzed (Participants) | 79
  DoublePI Therapy+Steroids/Alkylating Agent,>=4Line | 6.3
  Autologous transplant, Second Line: number analyzed (Participants) | 119
  Autologous transplant, Second Line | 2.5
  Autologous transplant, Third Line: number analyzed (Participants) | 71
  Autologous transplant, Third Line | 7.0
  Autologous transplant, Fourth Line or Later: number analyzed (Participants) | 85
  Autologous transplant, Fourth Line or Later | 1.2
  Allogeneic transplant, Second Line: number analyzed (Participants) | 119
  Allogeneic transplant, Second Line | 0.8
  Allogeneic transplant, Third Line: number analyzed (Participants) | 71
  Allogeneic transplant, Third Line | 1.4
  Allogeneic transplant, Fourth Line or Later: number analyzed (Participants) | 85
  Allogeneic transplant, Fourth Line or Later | 2.4
  Autologous or Allogeneic Transplant, Second Line: number analyzed (Participants) | 119
  Autologous or Allogeneic Transplant, Second Line | 2.5
  Autologous or Allogeneic Transplant, Third Line: number analyzed (Participants) | 71
  Autologous or Allogeneic Transplant, Third Line | 8.5
  Autologous or Allogeneic Transplant, >=4 Lines: number analyzed (Participants) | 85
  Autologous or Allogeneic Transplant, >=4 Lines | 3.5

4. Secondary Outcome: Percentage of MM Participants With Clinical and Sociodemographic Characteristics Categorized by Treatment Selection at the Latest Symptomatic Relapse and/or Refractory Episode
Description: Clinical and Sociodemographic variables categorized by treatment selection(immunomodulators[IMiDs],proteasome inhibitor[PI]+IMiDs,PI,monoclonal antibodies[mAb]): Age,sex(male/female),prior treatment lines(0,1,2,3 or more),prior relapses(0,1,2,3 or more),ISS disease stage(I:low risk,β2-Microglobulin<3.5mg/L,albumin≥3.5g/dL,II:not stage I or III,III:high risk,β2-Microglobulin≥5.5mg/L),CRAB signs(serum calcium>0.25mmol/L upper limit of normal,renal failure-creatinine clearance<40mL/min/serum creatinine>117μmol/L,anemia:reduction of hemoglobin(Hb)>2g/dL below lower limit of normal or Hb<10g/dL,bone lesions 1/more osteolytic lesion),risk according to cytogenetic profile(standard:trisomies,t[11;14];t[6;14];high:d[17p],t[14;16],t[14;20],other),other clinical variables:medullary/extramedullary plasmacytomas,osteopenia,fractures,neurological symptoms,infections,concomitant diseases:diabetes, neuropathy, COPD, cardiovascular disease, liver failure, psychiatric, neurological disorders.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
percentage of participants
  Age, 38-85 years, IMiDs: number analyzed (Participants) | 89
  Age, 38-85 years, IMiDs | 100
  Age, 43-76 years, PI + IMiDs: number analyzed (Participants) | 49
  Age, 43-76 years, PI + IMiDs | 100
  Age, 47-84 years, PI: number analyzed (Participants) | 34
  Age, 47-84 years, PI | 100
  Age, 39-80 years, mAb: number analyzed (Participants) | 61
  Age, 39-80 years, mAb | 100
  Age, 53-90 years, Other: number analyzed (Participants) | 26
  Age, 53-90 years, Other | 100
  Sex, Male, IMiDs: number analyzed (Participants) | 89
  Sex, Male, IMiDs | 49.4
  Sex, Female, IMiDs: number analyzed (Participants) | 89
  Sex, Female, IMiDs | 50.6
  Sex, Male, PI + IMiDs: number analyzed (Participants) | 49
  Sex, Male, PI + IMiDs | 61.2
  Sex, Female, PI + IMiDs: number analyzed (Participants) | 49
  Sex, Female, PI + IMiDs | 38.8
  Sex, Male, PI: number analyzed (Participants) | 34
  Sex, Male, PI | 47.1
  Sex, Female, PI: number analyzed (Participants) | 34
  Sex, Female, PI | 52.9
  Sex, Male, mAb: number analyzed (Participants) | 61
  Sex, Male, mAb | 55.7
  Sex, Female, mAb: number analyzed (Participants) | 61
  Sex, Female, mAb | 44.3
  Sex, Male, Other: number analyzed (Participants) | 26
  Sex, Male, Other | 57.7
  Sex, Female, Other: number analyzed (Participants) | 26
  Sex, Female, Other | 42.3
  Prior lines of treatment, 1, IMiDs: number analyzed (Participants) | 89
  Prior lines of treatment, 1, IMiDs | 50.6
  Prior lines of treatment, 2, IMiDs: number analyzed (Participants) | 89
  Prior lines of treatment, 2, IMiDs | 28.1
  Prior lines of treatment, 3 or more, IMiDs: number analyzed (Participants) | 89
  Prior lines of treatment, 3 or more, IMiDs | 21.3
  Prior lines of treatment, 1, PI + IMiDs: number analyzed (Participants) | 49
  Prior lines of treatment, 1, PI + IMiDs | 63.3
  Prior lines of treatment, 2, PI + IMiDs: number analyzed (Participants) | 49
  Prior lines of treatment, 2, PI + IMiDs | 16.3
  Prior lines of treatment, 3 or more, PI + IMiDs: number analyzed (Participants) | 49
  Prior lines of treatment, 3 or more, PI + IMiDs | 20.4
  Prior lines of treatment, 1, PI: number analyzed (Participants) | 34
  Prior lines of treatment, 1, PI | 44.1
  Prior lines of treatment, 2, PI: number analyzed (Participants) | 34
  Prior lines of treatment, 2, PI | 35.3
  Prior lines of treatment, 3 or more, PI: number analyzed (Participants) | 34
  Prior lines of treatment, 3 or more, PI | 20.6
  Prior lines of treatment, 1, mAb: number analyzed (Participants) | 61
  Prior lines of treatment, 1, mAb | 26.2
  Prior lines of treatment, 2, mAb: number analyzed (Participants) | 61
  Prior lines of treatment, 2, mAb | 29.5
  Prior lines of treatment, 3 or more, mAb: number analyzed (Participants) | 61
  Prior lines of treatment, 3 or more, mAb | 44.3
  Prior lines of treatment, 1, Other: number analyzed (Participants) | 26
  Prior lines of treatment, 1, Other | 11.5
  Prior lines of treatment, 2, Other: number analyzed (Participants) | 26
  Prior lines of treatment, 2, Other | 26.9
  Prior lines of treatment, 3 or more, Other: number analyzed (Participants) | 26
  Prior lines of treatment, 3 or more, Other | 61.5
  Number of prior relapses, 0, IMiDs: number analyzed (Participants) | 89
  Number of prior relapses, 0, IMiDs | 43.8
  Number of prior relapses, 1, IMiDs: number analyzed (Participants) | 89
  Number of prior relapses, 1, IMiDs | 31.5
  Number of prior relapses, 2, IMiDs: number analyzed (Participants) | 89
  Number of prior relapses, 2, IMiDs | 12.4
  Number of prior relapses, 3 and more, IMiDs: number analyzed (Participants) | 89
  Number of prior relapses, 3 and more, IMiDs | 12.4
  Number of prior relapses, 0, PI + IMiDs: number analyzed (Participants) | 49
  Number of prior relapses, 0, PI + IMiDs | 49.0
  Number of prior relapses, 1, PI + IMiDs: number analyzed (Participants) | 49
  Number of prior relapses, 1, PI + IMiDs | 36.7
  Number of prior relapses, 2, PI + IMiDs: number analyzed (Participants) | 49
  Number of prior relapses, 2, PI + IMiDs | 2.0
  Number of prior relapses, 3 or more, PI + IMiDs: number analyzed (Participants) | 49
  Number of prior relapses, 3 or more, PI + IMiDs | 12.2
  Number of prior relapses, 0, PI: number analyzed (Participants) | 34
  Number of prior relapses, 0, PI | 47.1
  Number of prior relapses, 1, PI: number analyzed (Participants) | 34
  Number of prior relapses, 1, PI | 32.4
  Number of prior relapses, 2, PI: number analyzed (Participants) | 34
  Number of prior relapses, 2, PI | 2.9
  Number of prior relapses, 3 or more, PI: number analyzed (Participants) | 34
  Number of prior relapses, 3 or more, PI | 17.6
  Number of prior relapses, 0, mAb: number analyzed (Participants) | 61
  Number of prior relapses, 0, mAb | 27.9
  Number of prior relapses, 1, mAb: number analyzed (Participants) | 61
  Number of prior relapses, 1, mAb | 26.2
  Number of prior relapses, 2, mAb: number analyzed (Participants) | 61
  Number of prior relapses, 2, mAb | 18.0
  Number of prior relapses, 3 or more, mAb: number analyzed (Participants) | 61
  Number of prior relapses, 3 or more, mAb | 27.9
  Number of prior relapses, 0, Other: number analyzed (Participants) | 26
  Number of prior relapses, 0, Other | 11.5
  Number of prior relapses, 1, Other: number analyzed (Participants) | 26
  Number of prior relapses, 1, Other | 26.9
  Number of prior relapses, 2, Other: number analyzed (Participants) | 26
  Number of prior relapses, 2, Other | 23.1
  Number of prior relapses, 3 or more, Other: number analyzed (Participants) | 26
  Number of prior relapses, 3 or more, Other | 38.5
  ISS Disease Stage I, IMiDs: number analyzed (Participants) | 65
  ISS Disease Stage I, IMiDs | 38.5
  ISS Disease Stage II, IMiDs: number analyzed (Participants) | 65
  ISS Disease Stage II, IMiDs | 38.5
  ISS Disease Stage III, IMiDs: number analyzed (Participants) | 65
  ISS Disease Stage III, IMiDs | 23.1
  ISS Disease Stage I, PI + IMiDs: number analyzed (Participants) | 39
  ISS Disease Stage I, PI + IMiDs | 51.3
  ISS Disease Stage II, PI + IMiDs: number analyzed (Participants) | 39
  ISS Disease Stage II, PI + IMiDs | 28.2
  ISS Disease Stage III, PI + IMiDs: number analyzed (Participants) | 39
  ISS Disease Stage III, PI + IMiDs | 20.5
  ISS Disease Stage I, PI: number analyzed (Participants) | 24
  ISS Disease Stage I, PI | 20.8
  ISS Disease Stage II, PI: number analyzed (Participants) | 24
  ISS Disease Stage II, PI | 54.2
  ISS Disease Stage III, PI: number analyzed (Participants) | 24
  ISS Disease Stage III, PI | 25.0
  ISS Disease Stage I, mAb: number analyzed (Participants) | 50
  ISS Disease Stage I, mAb | 40.0
  ISS Disease Stage II, mAb: number analyzed (Participants) | 50
  ISS Disease Stage II, mAb | 32.0
  ISS Disease Stage III, mAb: number analyzed (Participants) | 50
  ISS Disease Stage III, mAb | 28.0
  ISS Disease Stage I, Other: number analyzed (Participants) | 21
  ISS Disease Stage I, Other | 23.8
  ISS Disease Stage II, Other: number analyzed (Participants) | 21
  ISS Disease Stage II, Other | 23.8
  ISS Disease Stage III, Other: number analyzed (Participants) | 21
  ISS Disease Stage III, Other | 52.4
  CRAB Signs, None, IMiDs: number analyzed (Participants) | 89
  CRAB Signs, None, IMiDs | 29.2
  CRAB Signs, Some, IMiDs: number analyzed (Participants) | 89
  CRAB Signs, Some, IMiDs | 70.8
  CRAB Signs, None, PI + IMiDs: number analyzed (Participants) | 49
  CRAB Signs, None, PI + IMiDs | 14.3
  CRAB Signs, Some, PI + IMiDs: number analyzed (Participants) | 49
  CRAB Signs, Some, PI + IMiDs | 85.7
  CRAB Signs, None, PI: number analyzed (Participants) | 34
  CRAB Signs, None, PI | 20.6
  CRAB Signs, Some, PI: number analyzed (Participants) | 34
  CRAB Signs, Some, PI | 79.4
  CRAB Signs, None, mAb: number analyzed (Participants) | 61
  CRAB Signs, None, mAb | 31.1
  CRAB Signs, Some, mAb: number analyzed (Participants) | 61
  CRAB Signs, Some, mAb | 68.9
  CRAB Signs, None, Other: number analyzed (Participants) | 26
  CRAB Signs, None, Other | 23.1
  CRAB Signs, Some, Other: number analyzed (Participants) | 26
  CRAB Signs, Some, Other | 76.9
  Comorbidities, None, IMiDs: number analyzed (Participants) | 89
  Comorbidities, None, IMiDs | 41.6
  Comorbidities, Some, IMiDs: number analyzed (Participants) | 89
  Comorbidities, Some, IMiDs | 58.4
  Comorbidities, None, PI + IMiDs: number analyzed (Participants) | 49
  Comorbidities, None, PI + IMiDs | 49.0
  Comorbidities, Some, PI + IMiDs: number analyzed (Participants) | 49
  Comorbidities, Some, PI + IMiDs | 51.0
  Comorbidities, None, PI: number analyzed (Participants) | 34
  Comorbidities, None, PI | 35.3
  Comorbidities, Some, PI: number analyzed (Participants) | 34
  Comorbidities, Some, PI | 64.7
  Comorbidities, None, mAb: number analyzed (Participants) | 61
  Comorbidities, None, mAb | 32.8
  Comorbidities, Some, mAb: number analyzed (Participants) | 61
  Comorbidities, Some, mAb | 67.2
  Comorbidities, None, Other: number analyzed (Participants) | 26
  Comorbidities, None, Other | 23.1
  Comorbidities, Some, Other: number analyzed (Participants) | 26
  Comorbidities, Some, Other | 76.9
  Risk, High, IMiDs: number analyzed (Participants) | 10
  Risk, High, IMiDs | 50.0
  Risk, Standard, IMiDs: number analyzed (Participants) | 10
  Risk, Standard, IMiDs | 50.0
  Risk, High, PI + IMiDs: number analyzed (Participants) | 12
  Risk, High, PI + IMiDs | 41.7
  Risk, Standard, PI + IMiDs: number analyzed (Participants) | 12
  Risk, Standard, PI + IMiDs | 58.3
  Risk, High, PI: number analyzed (Participants) | 4
  Risk, High, PI | 50.0
  Risk, Standard, PI: number analyzed (Participants) | 4
  Risk, Standard, PI | 50.0
  Risk, High, mAb: number analyzed (Participants) | 15
  Risk, High, mAb | 60.0
  Risk, Standard, mAb: number analyzed (Participants) | 15
  Risk, Standard, mAb | 40.0
  Risk, High, Other: number analyzed (Participants) | 4
  Risk, High, Other | 50.0
  Risk, Standard, Other: number analyzed (Participants) | 4
  Risk, Standard, Other | 50.0
  Medullary Plasmacytoma, Yes, IMiDs: number analyzed (Participants) | 84
  Medullary Plasmacytoma, Yes, IMiDs | 15.5
  Medullary Plasmacytoma, No, IMiDs: number analyzed (Participants) | 84
  Medullary Plasmacytoma, No, IMiDs | 84.5
  Medullary Plasmacytoma, Yes, PI + IMiDs: number analyzed (Participants) | 44
  Medullary Plasmacytoma, Yes, PI + IMiDs | 25.0
  Medullary Plasmacytoma, No, PI + IMiDs: number analyzed (Participants) | 44
  Medullary Plasmacytoma, No, PI + IMiDs | 75.0
  Medullary Plasmacytoma, Yes, PI: number analyzed (Participants) | 34
  Medullary Plasmacytoma, Yes, PI | 14.7
  Medullary Plasmacytoma, No, PI: number analyzed (Participants) | 34
  Medullary Plasmacytoma, No, PI | 85.3
  Medullary Plasmacytoma, Yes, mAb: number analyzed (Participants) | 58
  Medullary Plasmacytoma, Yes, mAb | 8.6
  Medullary Plasmacytoma, No, mAb: number analyzed (Participants) | 58
  Medullary Plasmacytoma, No, mAb | 91.4
  Medullary Plasmacytoma, Yes, Other: number analyzed (Participants) | 25
  Medullary Plasmacytoma, Yes, Other | 16.0
  Medullary Plasmacytoma, No, Other: number analyzed (Participants) | 25
  Medullary Plasmacytoma, No, Other | 84.0
  Extramedullary Plasmacytoma, Yes, IMiDs: number analyzed (Participants) | 86
  Extramedullary Plasmacytoma, Yes, IMiDs | 12.8
  Extramedullary Plasmacytoma, No, IMiDs: number analyzed (Participants) | 86
  Extramedullary Plasmacytoma, No, IMiDs | 87.2
  Extramedullary Plasmacytoma, Yes, PI + IMiDs: number analyzed (Participants) | 48
  Extramedullary Plasmacytoma, Yes, PI + IMiDs | 33.3
  Extramedullary Plasmacytoma, No, PI + IMiDs: number analyzed (Participants) | 48
  Extramedullary Plasmacytoma, No, PI + IMiDs | 66.7
  Extramedullary Plasmacytoma, Yes, PI: number analyzed (Participants) | 34
  Extramedullary Plasmacytoma, Yes, PI | 11.8
  Extramedullary Plasmacytoma, No, PI: number analyzed (Participants) | 34
  Extramedullary Plasmacytoma, No, PI | 88.2
  Extramedullary Plasmacytoma, Yes, mAb: number analyzed (Participants) | 60
  Extramedullary Plasmacytoma, Yes, mAb | 6.7
  Extramedullary Plasmacytoma, No, mAb: number analyzed (Participants) | 60
  Extramedullary Plasmacytoma, No, mAb | 93.3
  Extramedullary Plasmacytoma, Yes, Other: number analyzed (Participants) | 25
  Extramedullary Plasmacytoma, Yes, Other | 24.0
  Extramedullary Plasmacytoma, No, Other: number analyzed (Participants) | 25
  Extramedullary Plasmacytoma, No, Other | 76.0
  Osteopenia, Yes, IMiDs: number analyzed (Participants) | 88
  Osteopenia, Yes, IMiDs | 23.9
  Osteopenia, No, IMiDs: number analyzed (Participants) | 88
  Osteopenia, No, IMiDs | 76.1
  Osteopenia, Yes, PI + IMiDs: number analyzed (Participants) | 48
  Osteopenia, Yes, PI + IMiDs | 6.3
  Osteopenia, No, PI + IMiDs: number analyzed (Participants) | 48
  Osteopenia, No, PI + IMiDs | 93.8
  Osteopenia, Yes, PI: number analyzed (Participants) | 34
  Osteopenia, Yes, PI | 8.8
  Osteopenia, No, PI: number analyzed (Participants) | 34
  Osteopenia, No, PI | 91.2
  Osteopenia, Yes, mAb: number analyzed (Participants) | 60
  Osteopenia, Yes, mAb | 13.3
  Osteopenia, No, mAb: number analyzed (Participants) | 60
  Osteopenia, No, mAb | 86.7
  Osteopenia, Yes, Other: number analyzed (Participants) | 26
  Osteopenia, Yes, Other | 23.1
  Osteopenia, No, Other: number analyzed (Participants) | 26
  Osteopenia, No, Other | 76.9
  Fractures, Yes, IMiDs: number analyzed (Participants) | 89
  Fractures, Yes, IMiDs | 15.7
  Fractures, No, IMiDs: number analyzed (Participants) | 89
  Fractures, No, IMiDs | 84.3
  Fractures, Yes, PI + IMiDs: number analyzed (Participants) | 49
  Fractures, Yes, PI + IMiDs | 18.4
  Fractures, No, PI + IMiDs: number analyzed (Participants) | 49
  Fractures, No, PI + IMiDs | 81.6
  Fractures, Yes, PI: number analyzed (Participants) | 34
  Fractures, Yes, PI | 11.8
  Fractures, No, PI: number analyzed (Participants) | 34
  Fractures, No, PI | 88.2
  Fractures, Yes, mAb: number analyzed (Participants) | 61
  Fractures, Yes, mAb | 14.8
  Fractures, No, mAb: number analyzed (Participants) | 61
  Fractures, No, mAb | 85.2
  Fractures, Yes, Other: number analyzed (Participants) | 26
  Fractures, Yes, Other | 15.4
  Fractures, No, Other: number analyzed (Participants) | 26
  Fractures, No, Other | 84.6
  Neurological Symptoms, Yes, IMiDs: number analyzed (Participants) | 89
  Neurological Symptoms, Yes, IMiDs | 10.1
  Neurological Symptoms, No, IMiDs: number analyzed (Participants) | 89
  Neurological Symptoms, No, IMiDs | 89.9
  Neurological Symptoms, Yes, PI + IMiDs: number analyzed (Participants) | 49
  Neurological Symptoms, Yes, PI + IMiDs | 10.2
  Neurological Symptoms, No, PI + IMiDs: number analyzed (Participants) | 49
  Neurological Symptoms, No, PI + IMiDs | 89.8
  Neurological Symptoms, Yes, PI: number analyzed (Participants) | 34
  Neurological Symptoms, Yes, PI | 5.9
  Neurological Symptoms, No, PI: number analyzed (Participants) | 34
  Neurological Symptoms, No, PI | 94.1
  Neurological Symptoms, Yes, mAb: number analyzed (Participants) | 61
  Neurological Symptoms, Yes, mAb | 1.6
  Neurological Symptoms, No, mAb: number analyzed (Participants) | 61
  Neurological Symptoms, No, mAb | 98.4
  Neurological Symptoms, Yes, Other: number analyzed (Participants) | 26
  Neurological Symptoms, Yes, Other | 11.5
  Neurological Symptoms, No, Other: number analyzed (Participants) | 26
  Neurological Symptoms, No, Other | 88.5
  MM Related Neurological Symptoms, Yes, IMiDs: number analyzed (Participants) | 89
  MM Related Neurological Symptoms, Yes, IMiDs | 5.6
  MM Related Neurological Symptoms, No, IMiDs: number analyzed (Participants) | 89
  MM Related Neurological Symptoms, No, IMiDs | 94.4
  MM Related Neurological Symptoms, Yes, PI + IMiDs: number analyzed (Participants) | 49
  MM Related Neurological Symptoms, Yes, PI + IMiDs | 8.2
  MM Related Neurological Symptoms, No, PI + IMiDs: number analyzed (Participants) | 49
  MM Related Neurological Symptoms, No, PI + IMiDs | 91.8
  MM Related Neurological Symptoms, Yes, PI: number analyzed (Participants) | 34
  MM Related Neurological Symptoms, Yes, PI | 5.9
  MM Related Neurological Symptoms, No, PI: number analyzed (Participants) | 34
  MM Related Neurological Symptoms, No, PI | 94.1
  MM Related Neurological Symptoms, Yes, mAb: number analyzed (Participants) | 61
  MM Related Neurological Symptoms, Yes, mAb | 0.0
  MM Related Neurological Symptoms, No, mAb: number analyzed (Participants) | 61
  MM Related Neurological Symptoms, No, mAb | 100.0
  MM Related Neurological Symptoms, Yes, Other: number analyzed (Participants) | 26
  MM Related Neurological Symptoms, Yes, Other | 7.7
  MM Related Neurological Symptoms, No, Other: number analyzed (Participants) | 26
  MM Related Neurological Symptoms, No, Other | 92.3
  Infections, Yes, IMiDs: number analyzed (Participants) | 89
  Infections, Yes, IMiDs | 14.6
  Infections, No, IMiDs: number analyzed (Participants) | 89
  Infections, No, IMiDs | 85.4
  Infections, Yes, PI + IMiDs: number analyzed (Participants) | 49
  Infections, Yes, PI + IMiDs | 20.4
  Infections, No, PI + IMiDs: number analyzed (Participants) | 49
  Infections, No, PI + IMiDs | 79.6
  Infections, Yes, PI: number analyzed (Participants) | 34
  Infections, Yes, PI | 14.7
  Infections, No, PI: number analyzed (Participants) | 34
  Infections, No, PI | 85.3
  Infections, Yes, mAb: number analyzed (Participants) | 61
  Infections, Yes, mAb | 11.5
  Infections, No, mAb: number analyzed (Participants) | 61
  Infections, No, mAb | 88.5
  Infections, Yes, Other: number analyzed (Participants) | 26
  Infections, Yes, Other | 11.5
  Infections, No, Other: number analyzed (Participants) | 26
  Infections, No, Other | 88.5

5. Secondary Outcome: Number of New Relevant Variables That Are Not Currently Collected in Clinical Records and That Could Influence in the Disease Management at Relapse
Time Frame: Day 1
Population: Data was not collected for this outcome measure.
Units Other Than Participants: Variables
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 0
Number analyzed (Variables) | 0

6. Secondary Outcome: Health-Related Quality of Life (HRQOL) Based on European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire- Core 30
Description: The EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale. Most of the 30 items have 4 response levels (not at all, a little, quite a bit, and very much), with 2 questions relying on a 7-point numeric rating scale with a recall period of the previous week. Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QOL scale, higher scores represent better QOL; for the symptom scales, lower scores represent better QOL.
Time Frame: Day 1
Population: All participants eligible for analyses were included. Overall number of participants analyzed are the participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 273
score on a scale | 53.5 (23.9)

7. Secondary Outcome: HRQOL Based on EORTC Multiple Myeloma Module (EORTC QLQ-MY20) Subscale Score
Description: The EORTC QLQ-MY20 has 20 items across 4 independent subscales, 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms, and side effects of treatment) with a recall period of previous week. Scores from each subscale were transformed from 0 to 100. For the functional scales, high scores represent improvement. For the symptom scales, higher scores represent worsening.
Time Frame: Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 273
score on scale
  Future perspective | 58.4 (27.7)
  Body image | 72.9 (34.4)
  Symptoms of the disease | 30.7 (23.2)
  Adverse effects of the treatment | 25.4 (17.2)

8. Secondary Outcome: HRQOL Based on the Spanish Translated Version of EORTC Multiple Myeloma Module (EORTC QLQ-MY20)
Description: The EORTC QLQ-MY20 has 20 items across 4 independent subscales, 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms, and side effects of treatment) with a recall period of previous week. Scores from each subscale were transformed from 0 to 100. For the functional scales, high scores represent improvement. For the symptom scales, higher scores represent worsening. Spanish Translated Version of EORTC Multiple Myeloma Module included 4 factors, each factor corresponds to questions related to the particular component of the scale. Factor I indicate symptoms. Factor II indicates future perspectives. Factor III indicate adverse effects of the treatment. Factor IV indicates adverse effects of the treatment and body image. Each of these factors were used for the clinical validity of the scale.
Time Frame: Day 1
Population: All participants eligible for analyses were included. Number analyzed is the number of participants with data available for analyses for the specific category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
score on a scale
  Future perspective, Factors I-II: number analyzed (Participants) | 142
  Future perspective, Factors I-II | 60.3 (28.2)
  Future perspective, Factors III: number analyzed (Participants) | 53
  Future perspective, Factors III | 53.9 (24.9)
  Body image, Factors I-II: number analyzed (Participants) | 142
  Body image, Factors I-II | 73.9 (35.5)
  Body image, Factors III: number analyzed (Participants) | 53
  Body image, Factors III | 73.0 (32.7)
  Symptoms of the disease, Factors I-II: number analyzed (Participants) | 142
  Symptoms of the disease, Factors I-II | 31.9 (23.6)
  Symptoms of the disease, Factors III: number analyzed (Participants) | 53
  Symptoms of the disease, Factors III | 27.3 (22.1)
  Adverse effects of the treatment, Factors I-II: number analyzed (Participants) | 142
  Adverse effects of the treatment, Factors I-II | 24.3 (16.9)
  Adverse effects of the treatment, Factors III: number analyzed (Participants) | 53
  Adverse effects of the treatment, Factors III | 29.0 (17.5)

9. Secondary Outcome: Percentage of Participants With Health Care Resource Utilization (HU)
Description: Healthcare resources used during medical encounters include intensive care unit (ICU) admissions, hospital admissions, visits to the emergency room, days admitted.
Time Frame: Day 1
Population: All participants eligible for analyses were included.
Measure: Number; unit: percentage of participants
Arm/Group | Multiple Myeloma (MM) Participants
Number analyzed (Participants) | 276
percentage of participants
  Admitted at some healthcare service | 56.2
  Admitted to Hospital | 59.4
  Used ambulance to attend to the hospital | 7.0
  Used their own transport | 67.8
  Consultation with the primary care physician | 21.7
  Consultation with the oncologist | 2.5
  Consultation with the psychologist | 3.6
  Attended psychologist | 60
  Attended hematologist | 89.1
  Required some test | 82.2
  Had undergone X-ray test | 43.2

ADVERSE EVENTS:
Time Frame: From enrollment on 26 July 2017 to last date of assessment 30 January 2019 (Up to 1.5 years)
Description: Data of adverse events or adverse drug reactions were not collected as part of the study database.
Arm/Group | Multiple Myeloma (MM) Participants
All-Cause Mortality (participants affected / at risk) | 0/276
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03188536/Prot_SAP_000.pdf